CLINICAL TRIAL: NCT06485622
Title: Outcome and Improvement of Different Treatment in Arteriosclerosis Obliterans: a Prospective, Single-center, Observational Study
Brief Title: Outcome and Improvement of Different Treatment in Arteriosclerosis Obliterans
Status: Recruiting | Type: Observational
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Zilun Li, Clinical Professor, First Affiliated Hospital, Sun Yat-Sen University
Other Study IDs: [2024]225
Record Dates: First submitted 2024-06-20; First posted 2024-07-03 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Arteriosclerosis Obliterans
MeSH Terms: conditions — Arteriosclerosis Obliterans

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (6):
- Bypass group: open bypass group
  Interventions: Procedure: open bypass group
- BMS group: BMS (bare metal stent) group
  Interventions: Procedure: bare metal stent group
- POBA group: POBA (plain old balloon angioplasty) group
  Interventions: Procedure: plain old balloon angioplasty group
- DCB group: drug-coated balloon group
  Interventions: Procedure: drug-coated balloon group
- DA group: DA (directional atherectomy) group
  Interventions: Procedure: directional atherectomy group
- HR group: HR (hybrid repair) group
  Interventions: Procedure: hybrid repair group

INTERVENTIONS:
Procedure: open bypass group — After heparinization, the target artery is clamped above and below the anastomosis. The target artery is dissected along the anterior wall, calcium portions or mural thrombus are removed. Graft (autologous or prosthetic graft) is cut obliquely and anastomosis suturing starts with distal angle. Next stage is tunnel creating for graft conduction.
  Groups: Bypass group
Procedure: bare metal stent group — Bare metal stent implantation during the index procedure.
  Groups: BMS group
Procedure: plain old balloon angioplasty group — Only plain old balloon was used during the index procedure.
  Groups: POBA group
Procedure: drug-coated balloon group — Drug-coated balloon was used during the index procedure.
  Groups: DCB group
Procedure: directional atherectomy group — Directional atherectomy (with or without drug-coated balloon) during the index procedure.
  Groups: DA group
Procedure: hybrid repair group — Femoral artery arteriotomy. Further execute a direct endarterectomy femoral artery and from the mouth of a hip artery. Arteriotomy of the femoral artery is closed with a vascular patch use (synthetic or biological). Endovascular revascularization followed.
  Groups: HR group

SUMMARY:
This study is a prospective, single-center, observational study. In this study, we aim to evaluate the clinical outcome and cost-effectiveness of different treatments of lower extremity arterial occlusive disease. It is expected to include about 400 patients diagnosed with lower extremity arterial occlusive disease in our center from July 2024 to July 2026. All enrolled patients will be followed for three years. All patients diagnosed with arteriosclerosis obliterans (ASO) and all treatment techniques were included in this study. The primary outcomes include the Efficacy and Safety End Points of each techniques.

DETAILED DESCRIPTION:
Arteriosclerosis obliterans (ASO) is a kind of lower extremity arterial disease which occurs frequently in middle-aged and elderly people. The incidence of ASO increases with age. In patients with ASO, the build-up of fatty deposits, cholesterol, and other substances (plaques) in the arteries reduces blood flow to the extremities. This can lead to symptoms such as leg pain, cramping, and fatigue, especially during physical activity. In severe cases, it may result in pain at rest, non-healing wounds, and complications such as tissue damage or infection. Chronic wound is one of the symptoms that affect the quality of life. Therefore, wound healing is also an important index for postoperative care. However, no study has reported detailed performance data for different treatments. As an auxiliary method in clinical treatment, nutrition plays an important role in improving the clinical outcome of patients in the development and postoperative stages of the disease. The effect of nutritional risk assessment and nutritional education on postoperative symptoms of ASO has not been reported. Therefore, we plan to carry out this prospective, single-center, observational study, providing new data on the efficacy, safety and cost-effectiveness for different treatment and assistive techniques in lower extremity arterial occlusive disease.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older, gender is not limited.
2. Patients diagnosed with arteriosclerosis obliterans.
3. Rutherford stages 2-6.
4. When there are multiple stenosis lesions, the treatment of the most severe lesion is included.
5. Patients with at least one arterial occlusion ( iliac, femoral, popliteal, anterior tibial, posterior tibial, and/or peroneal artery) of the lower extremity were included.

Exclusion Criteria:

1. Malignant tumor
2. Alzheimer's disease
3. Blood disease or bleeding tendency
4. Heart Failure Grade III ~ IV
5. Pregnancy or lactation
6. An above-knee-below-knee amputation has been performed
7. Unable to accept therapeutic function tests
8. Life expectancy is less than six months
9. Combined with other diseases affecting walking
10. Cardiovascular and cerebrovascular events occurred within 3 months, including non-fatal myocardial infarction, unstable angina, stable angina, non-fatal ischemic stroke and hemorrhagic stroke
11. Patients with significant abnormal liver and renal function that the investigators judged to be clinically significant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: lower extremity arteriosclerosis obliterans
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
Limb salvage rate | 1 month; 6 months; 12 months; 24 months; 36 months
  Freedom from above ankle amputation in target limb.
Primary patency rate | 1 month; 6 months; 12 months; 24 months; 36 months
  Primary patency of target lesion is assessed by the vascular ultrasound.
Major adverse limb event (MALE) rate | 1 month; 6 months; 12 months; 24 months; 36 months
  Major adverse limb events include anyone of the following: Amputation in target limb and major re-intervention on target limb.
All cause mortality rate | 1 month; 6 months; 12 months; 24 months; 36 months
  Death due to any cause.

SECONDARY OUTCOMES:
Restenosis of the target lesion | 1 month; 6 months; 12 months; 24 months; 36 months
  A peak systolic velocity ratio of over 2.4 measured using duplex ultrasound, >50% diameter stenosis or occlusion by follow-up angiography.
Major adverse cardiovascular events (MACE) | 1 month; 6 months; 12 months; 24 months; 36 months
  Major adverse cardiovascular events include anyone of the following: Major amputations, myocardial infarction, ischemic stroke, arterial puncture problems requiring intervention, and acute kidney failure associated with endovascular therapy.
Quality-adjusted life-years (QALYs) | 1 month; 6 months; 12 months; 24 months; 36 months
  Time is measured in years and the VascuQol (Vascular Quality-of-Life, scored on a scale from 1 to 7 by using the VascuQol-25 questionnaire) on an index scale ranging from 1 (worst possible) to 7(best possible). The total number of QALYs was calculated by multiplying the HRQoL index score (QALY weight) by the time spent in each health state. One QALY can be viewed as living for 1 year in the best possible health.
Survival Rate | 1 month; 6 months; 12 months; 24 months; 36 months
  Telephone follow-up visit and/or medical chart review and/or publicly available records consultation for vital status.

OTHER OUTCOMES:
Clinically-driven target lesion revascularization (CD-TLR) | 1 month; 6 months; 12 months; 24 months; 36 months
  Any surgical or percutaneous intervention to the target lesion(s) after the index procedure.
Wound healing | 1 month; 6 months; 12 months; 24 months; 36 months
  The wound diameter and ulcer grade.
Incremental cost effectiveness ratio (ICER) | 1 month; 6 months; 12 months; 24 months; 36 months
  The difference in costs are divided by the difference in QALY or VascuQol.
Improvement of dietary and life style | 1 month; 6 months; 12 months; 24 months; 36 months
  The dietary habits and lifestyle of the patients were collected by questionnaire before operation. Before discharge, patients received education on healthy diet and lifestyle, and information on diet and lifestyle was collected at follow-up.
Cost effectiveness acceptability curve | 1 month; 6 months; 12 months; 24 months; 36 months
  It shows the probability of one treatment being more efficient in terms of QALYs than the other treatment for different levels of willingness to pay.
Ankle brachial index (ABI) | 1 month; 6 months; 12 months; 24 months; 36 months
  The ratio of systolic pressure measured at the ankle artery to the brachial artery.

CONTACTS AND LOCATIONS:
Overall Officials: Zilun Li, Principal Investigator — First Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Scully RE, Arnaoutakis DJ, DeBord Smith A, Semel M, Nguyen LL. Estimated annual health care expenditures in individuals with peripheral arterial disease. J Vasc Surg. 2018 Feb;67(2):558-567. doi: 10.1016/j.jvs.2017.06.102. Epub 2017 Aug 25. PMID 28847660
- [Background] Fowkes FG, Aboyans V, Fowkes FJ, McDermott MM, Sampson UK, Criqui MH. Peripheral artery disease: epidemiology and global perspectives. Nat Rev Cardiol. 2017 Mar;14(3):156-170. doi: 10.1038/nrcardio.2016.179. Epub 2016 Nov 17. PMID 27853158
- [Background] Soga Y, Iida O, Takahara M, Hirano K, Suzuki K, Kawasaki D, Miyashita Y, Tsuchiya T. Two-year life expectancy in patients with critical limb ischemia. JACC Cardiovasc Interv. 2014 Dec;7(12):1444-9. doi: 10.1016/j.jcin.2014.06.018. PMID 25523536
- [Background] Gupta R, Siada S, Lai S, Al-Musawi M, Malgor EA, Jacobs DL, Malgor RD. Critical appraisal of the contemporary use of atherectomy to treat femoropopliteal atherosclerotic disease. J Vasc Surg. 2022 Feb;75(2):697-708.e9. doi: 10.1016/j.jvs.2021.07.106. Epub 2021 Jul 22. PMID 34303802
- [Background] Fu S, Zhao H, Shi J, Abzhanov A, Crawford K, Ohno-Machado L, Zhou J, Du Y, Kuo WP, Zhang J, Jiang M, Jin JG. Peripheral arterial occlusive disease: global gene expression analyses suggest a major role for immune and inflammatory responses. BMC Genomics. 2008 Aug 1;9:369. doi: 10.1186/1471-2164-9-369. PMID 18673543
- [Background] Folkersen L, Persson J, Ekstrand J, Agardh HE, Hansson GK, Gabrielsen A, Hedin U, Paulsson-Berne G. Prediction of ischemic events on the basis of transcriptomic and genomic profiling in patients undergoing carotid endarterectomy. Mol Med. 2012 May 9;18(1):669-75. doi: 10.2119/molmed.2011.00479. PMID 22371308